CLINICAL TRIAL: NCT00426907
Title: Weightbearing After Proximal Open-wedge Tibial Osteotomy - a Clinical, Randomized RSA-study.
Brief Title: Weightbearing After High Tibial Osteotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON-04-016-TLH
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Osteotomy; Healing; Rehabilitation; Roentgen Stereometric Analysis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Full postoperative weightbearing
  Interventions: Procedure: Unlimited postoperative weightbearing
- 2 (Active Comparator): Partial weightbearing 6 weeks postoperative
  Interventions: Procedure: Unlimited postoperative weightbearing

INTERVENTIONS:
Procedure: Unlimited postoperative weightbearing — Unlimited postoperative weightbearing

SUMMARY:
In this project we want investigate the clinical results after different rehabilitation regimens(Limited or unlimited weightbearing after surgery) in Open-wedge High Tibial Osteotomies.

The hypothesis is that unlimited weightbearing is beneficial for the healing and rehabilitation.

DETAILED DESCRIPTION:
In the treatment of osteoarthritis of the medial compartment of the knee, Open wedge high tibial osteotomy is a good choice of treatment for the young and active patient.

However it leaves an open gap which has to be filled with a bone substitute and requires stable fixation.

Different rehabilitation-regimens are described, many advocating a period of partial weight-bearing for a period after surgery.

Results from biomechanical studies suggest that immediate full weight-bearing is safe, enabling earlier mobilisation without compromising safe solid healing.

The aim of the present study is to evaluate whether there is any difference in clinical outcome, correction, stability and healing in open-wedge osteotomies (osteosynthesis with the Dynafix® system (EBI)) after 2 different rehabilitation regimens: Limited weight-bearing (20 kg) for 6 weeks, and unrestricted weight-bearing.

The investigation is performed as a randomised prospective clinical trial including 20 patients with a planned 2 years follow-up period.

Clinical outcome is evaluated with: Hospital of special surgery score, KOOS, SF 12 and Lysholm score.

Routine standing x-rays is performed. Stability of the osteotomy is assessed with Roentgen Stereophotogrammetric Analysis (RSA) that provides the opportunity of exact 3-dimensional measuring of eventual loss of correction.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Osteoarthritis of medial compartment of the knee, Ahlbäck gr. 1-2
* Varus deformity

Exclusion Criteria:

* Prednisolone treatment.
* NSAID treatment.
* BMI > or = 35.
* Previous surgery in lateral knee compartment.
* Secondary Arthrosis following fracture(s) of the tibial condyle(s).
* Lack of informed consent.
* Correction >12,5 mm
* Peroperative displaced fracture of lateral bony hinge.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Migration in mm measured with RSA (Roentgen Stereometric Analysis): | Postoperative, at 3 month, 1 and 2 years.

SECONDARY OUTCOMES:
Clinical scores including range of Movement and muscular status at 6 weeks, 3 month, 1 and 2 years postoperative. | Postoperative, at 3 month, 1 and 2 years.
Hip-Knee-Ankle axis at 3 month, 1 and 2 years postoperative. | Postoperative, at 3 month, 1 and 2 years.
Bone Mineral Density (DEXA-scan) pre-op., Post.-op, at 6 weeks, 3 months and 1 and 2 years postop. | Postoperative, at 3 month, 1 and 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lind-Hansen, MD, Principal Investigator — Orthopaedic Division, Northern Denmark Region
Locations (1):
- Northern Orthopaedic Division, Klinik Farsoe and Aarhus University Hospital, Farsø, Northern Jutland, Denmark